CLINICAL TRIAL: NCT04118660
Title: Thoracic Specimen Registry
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Eric S. Edell, Prinicpal, Mayo Clinic
Other Study IDs: 16-009655
Record Dates: First submitted 2019-01-07; First posted 2019-10-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Thoracic Diseases; Lung Cancer; Lung Transplant
MeSH Terms: conditions — Thoracic Diseases; Lung Neoplasms | interventions — Tissue Banks

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Biospecimen Retention: Samples With DNA — A blood sample will be collected at the time of consent/baseline. Optional subsequent blood draws maybe requested no more frequently than every 8 weeks. Patients scheduled for their clinically indicated thoracic procedure and have excess of clinical diagnostic tissue available will have tissue kept in the registry for future research. Patients scheduled for their clinical indicated bronchoscopy or CT guided procedure may have a sample go through the Touch Prep process and slides/cells will be kept for future research.
  Patients scheduled for clinically indicated bronchoscopy with bronchoalveolar lavage BAL or Thoracentesis (TAP) procedure as part of that procedure may have fluid that is in excess of clinical diagnostic material, saved of future research. In addition, at the time of any future clinically indicated blood draws, thoracic procedures, thoracic resections, or metastatic thoracic primary tumors resections from other organs tissue will be requested for the research study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thoracic Disease: Thoracic Diseases (which includes but not limited to the following: thoracic neoplasms (masses/nodules) malignant or benign, interstitial lung diseases (ILD), chronic obstructive pulmonary disease (COPD), thoracic infections, thoracic malignancies metastatic to other organs, other cancers metastatic to the thoracic cavity.
  Interventions: Other: Tissue Banking

INTERVENTIONS:
Other: Tissue Banking — Blood, tissue, and fluid collection

SUMMARY:
The purpose of the registry will be to support ongoing research in the etiology, early diagnosis, clinical management, and prognosis of lung cancer and other cancers and diseases of the thorax by developing a complete repository of specimens from patients with thoracic disease including but not limited to suspected lung cancer, mediastinal and pleural tumors, lung transplants and from patients at a very high risk of developing other thoracic cancers or other thoracic diseases.

DETAILED DESCRIPTION:
The primary objective of this proposal is to develop a Thoracic Specimen Registry at Mayo Clinic. The purpose of the registry will be to support ongoing research in the etiology, early diagnosis, clinical management, and prognosis of lung cancer and other cancers and diseases of the thorax by developing a complete repository of specimens from patients with thoracic disease including but not limited to suspected lung cancer, mediastinal and pleural tumors, lung transplants and from patients at a very high risk of developing other thoracic cancers or other thoracic diseases. Collected specimens will include peripheral blood, bronchoalveolar lavage (BAL) fluid, pleural fluid, tissue (surgical resections & biopsies) and touch prep samples. The specimens will be stored in a central location at Mayo Clinic and managed by the Mayo Clinic Thoracic Specimen Registry Steering Committee. The registry will be a foundation for the development and implementation of research protocols and clinical trials that will enhance current knowledge of etiology and detection, discovery of new molecular and biochemical markers for screening, early diagnosis, and develop state-of-the-art therapeutic and preventive interventions for managing patients with, or at risk for, thoracic cancers or other thoracic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be > 18 years of age
* Presumed or known or screening of Thoracic Diseases (which includes but not limited to the following: thoracic neoplasms (masses/nodules) malignant or benign, interstitial lung diseases (ILD), chronic obstructive pulmonary disease (COPD), thoracic infections, thoracic malignancies metastatic to other organs, other cancers metastatic to the thoracic cavity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic Rochester patients with thoracic disease
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Thoracic Specimen Repository | Through study completion, approximately 10 years
  Number of thoracic specimens collected

CONTACTS AND LOCATIONS:
Overall Officials: Eric Edell, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials